CLINICAL TRIAL: NCT03764020
Title: A Triple Blinded Randomized Controlled Trial of Oral Melatonin in Elevated Blood Pressure Individual (MRCTEBP)
Brief Title: Trial of Oral Melatonin in Elevated Blood Pressure
Acronym: MRCTEBP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zinat Hatmi, Professor, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TUMS
Record Dates: First submitted 2018-11-27; First posted 2018-12-04 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Elevated Blood Pressure
Keywords: melatonin; inflammatory biomarkers
MeSH Terms: conditions — Hypertension | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Melatonin 3 Mg or placebo associated with life style modification according to 2013ACC/ AHA guideline has been planned in parallel fashion for three weeks of follow up. Participants allocated to each group will stay at the same interventional group for entire follow up period of three weeks.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Triple blinding is planned. All participants, medical providers and outcome evaluators will be blinded about treatment arms.
  The THC pharmacy will dispense the medication and perform the randomization. Melatonin capsule and placebo will be completely identical.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin (Experimental): Intervention group1:
  Melatonin,capsule,3 mg, one dose one hour before bedtime, three weeks
  Interventions: Drug: Melatonin/experimental
- Placebo (Placebo Comparator): Intervention group2 :
  Placebo, capsule, 3 mg, one dose one hour before bedtime, for three weeks
  Interventions: Drug: Placebo oral capsule/placebo comparator

INTERVENTIONS:
Drug: Placebo oral capsule/placebo comparator — 3 mg placebo capsule one hour before bedtime for three weeks along with life style modification according to ACC/AHA 2013 guideline
  Other Names: Placebo
  Arms: Placebo
Drug: Melatonin/experimental — Melatonin ,capsule, 3 mg, one dose one hour before bedtime, for three weeks along with life style modification according to ACC/AHA 2013 guideline.
  Other Names: Melatona
  Arms: Melatonin

SUMMARY:
Since, lowering blood pressure (BP) in elevated blood pressure individuals represents an excellent opportunity to for primary prevention of hypertension (HTN). Therefore, it is planned to use a safe treatment option - oral melatonin supplementation - associated with lifestyle interventions according to the American college of cardiology/American heart association (ACC/AHA) 2013 guideline in elevated blood pressure individuals to mitigate systolic and diastolic BP and ultimately, to prevent the development of HTN.

Hypothesis:

Melatonin therapy can lower the systolic and diastolic BP of elevated blood pressure individuals Melatonin can attenuate levels of circulatory biomarkers of Hs- CRP, Cholesterol, LDL-c and triglyceride

DETAILED DESCRIPTION:
Study design: Randomized controlled trial (RCT)

Study population: Elevated blood pressure individuals who present themselves at the outpatient clinics of Tehran Heart Centre(THC) , seeking blood pressure treatment and who have a systolic blood pressure of 120-129 mmHg or a diastolic blood pressure of =80 mmHg.

Treatment groups: Melatonin 3 mg versus placebo

sample size: 160 per group ( 320 overall)

Treatment allocation: After completing informed consent and prior to randomization, all participants undergo complete physical examination and laboratory test. Baseline levels of inflammatory biomarkers and pregnancy test (for women in reproductive age) will be performed. Sleep quality, actual sleep time, and sleep latency will be recorded.

Treatment plan: Three weeks melatonin 3 Mg or placebo one hour before bedtime has been planned. All of the melatonin and placebo capsules will be supplied from a single hospital pharmacy and free of charge to the participants. Melatonin and placebo capsules will be identical. Participants will receive a three weeks supply at the assignment time. Besides, all participants will receive a careful plan of adherence to a heart-healthy diet, regular exercise, instruction for avoidance of tobacco use and maintenance of a healthy body mass index (BMI) according to 2013ACC/ AHA guideline.

Follow up: Three weeks

ELIGIBILITY:
Inclusion Criteria:

* Individuals with systolic blood pressure120-129 and/or diastolic blood pressure =80mmHg
* Negative pregnancy test for women at productive age
* Baseline melatonin and biomarkers level and complete liver function tests within normal range

Exclusion Criteria:

* Previous history of hypersensitivity of melatonin
* Past history of using antihypertensive treatment
* Past medical history of hypertension, cardiovascular diseases, (i.e. coronary artery disease), and diabetes mellitus, epilepsy and other physician documented diseases
* Use of beta-blockers, sleep aids, warfarin, flaxseed, soy and supplements

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 320 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Mean change in systolic blood pressure from baseline | From enrollment to end of treatment at 3 weeks
  Mean change in Systolic blood pressure from baseline in Millimeter Mercury, it measures average changes in systolic blood pressure. The best outcome value is < and =120 millimeter mercury. Systolic blood pressure ranges between 90-250 millimeter mercury.
Mean change in diastolic blood pressure from baseline | From enrollment to end of treatment at 3 weeks
  Mean change in diastolic blood pressure from baseline in Millimeter Mercury, it measures average changes in systolic blood pressure. The best outcome value is < 80 millimeter mercury. Diastolic blood pressure ranges between 60-140 millimeter mercury.
Mean change in cholesterol | From enrollment to end of treatment at 3 weeks
  Mean change in cholesterol in Milligram/deciliter from baseline, it measures average changes in cholesterol. The best outcome value is 200 milligram per deciliter. Total cholesterol less than 200 milligram per deciliter are considered desirable for adults. A reading between200-239 is considered borderline and a reading of 240 above is considered high.
Mean change in low density lipoprotein | From enrollment to end of treatment at 3 weeks
  Mean change in low density lipoprotein in Milligram/deciliter from baseline, it measures average changes in low density lipoprotein. The best outcome value is 100 milligram per deciliter. LDL level less than 100 milligram per deciliter is considered desirable, 100-130 borderline, 130-189 borderline high and above 190 is considered high.
Mean change in fasting blood sugar | From enrollment to end of treatment at 3 weeks
  Mean change in fasting blood sugar in Milligram/deciliter from baseline, it measures average changes in fasting blood sugar. Fasting blood sugar 72-99 milligram per deciliter is considered normal, 100-116 borderline and above 116 is considered high.
Mean change in inflammatory biomarker | From enrollment to end of treatment at 3 weeks
  Mean change in high sensitive C reactive protein (Hs-CRP) in Milligram/liter, it measures average changes in high sensitive C reactive protein (Hs-CRP). The best outcome value is <= 3 milligram per liter.
  1-3 milligram per liter is considered normal and above 3 is considered high.

SECONDARY OUTCOMES:
Mean change in sleep quality score from baseline | From enrollment to end of treatment at 3 weeks
  Mean change in Pittsburg sleep quality questionnaire in Likert numerical score from baseline, it measures average changes in sleep quality score. Pittsburg sleep quality questionnaire score of 5 or greater is indicative of poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: zinat Hatmi, Dr, Principal Investigator — Tehran University of Medical Sciences

IPD SHARING:
Plan to Share IPD: Undecided
In case of designing systematic reviews and according to Helsinki declaration might be shared.

REFERENCES:
- [Background] Ekmekcioglu C, Thalhammer T, Humpeler S, Mehrabi MR, Glogar HD, Holzenbein T, Markovic O, Leibetseder VJ, Strauss-Blasche G, Marktl W. The melatonin receptor subtype MT2 is present in the human cardiovascular system. J Pineal Res. 2003 Aug;35(1):40-4. doi: 10.1034/j.1600-079x.2003.00051.x. PMID 12823612
- [Background] Hardeland R, Cardinali DP, Srinivasan V, Spence DW, Brown GM, Pandi-Perumal SR. Melatonin--a pleiotropic, orchestrating regulator molecule. Prog Neurobiol. 2011 Mar;93(3):350-84. doi: 10.1016/j.pneurobio.2010.12.004. Epub 2010 Dec 28. PMID 21193011
- [Background] Jonas M, Garfinkel D, Zisapel N, Laudon M, Grossman E. Impaired nocturnal melatonin secretion in non-dipper hypertensive patients. Blood Press. 2003;12(1):19-24. PMID 12699131
- [Background] Girotti L, Lago M, Ianovsky O, Elizari MV, Dini A, Perez Lloret S, Albornoz LE, Cardinali DP. Low urinary 6-sulfatoxymelatonin levels in patients with severe congestive heart failure. Endocrine. 2003 Dec;22(3):245-8. doi: 10.1385/ENDO:22:3:245. PMID 14709797
- [Background] Dominguez-Rodriguez A, Abreu-Gonzalez P, Garcia MJ, Sanchez J, Marrero F, de Armas-Trujillo D. Decreased nocturnal melatonin levels during acute myocardial infarction. J Pineal Res. 2002 Nov;33(4):248-52. doi: 10.1034/j.1600-079x.2002.02938.x. PMID 12390508
- [Background] Dominguez-Rodriguez A, Abreu-Gonzalez P, Sanchez-Sanchez JJ, Kaski JC, Reiter RJ. Melatonin and circadian biology in human cardiovascular disease. J Pineal Res. 2010 Aug;49(1):14-22. doi: 10.1111/j.1600-079X.2010.00773.x. Epub 2010 Jun 1. PMID 20536686
- [Background] Arangino S, Cagnacci A, Angiolucci M, Vacca AM, Longu G, Volpe A, Melis GB. Effects of melatonin on vascular reactivity, catecholamine levels, and blood pressure in healthy men. Am J Cardiol. 1999 May 1;83(9):1417-9. doi: 10.1016/s0002-9149(99)00112-5. PMID 10235107
- [Background] Cagnacci A, Arangino S, Angiolucci M, Maschio E, Longu G, Melis GB. Potentially beneficial cardiovascular effects of melatonin administration in women. J Pineal Res. 1997 Jan;22(1):16-9. doi: 10.1111/j.1600-079x.1997.tb00297.x. PMID 9062865
- [Background] Cagnacci A, Arangino S, Angiolucci M, Maschio E, Melis GB. Influences of melatonin administration on the circulation of women. Am J Physiol. 1998 Feb;274(2):R335-8. doi: 10.1152/ajpregu.1998.274.2.R335. PMID 9486289
- [Background] Scheer FA, Van Montfrans GA, van Someren EJ, Mairuhu G, Buijs RM. Daily nighttime melatonin reduces blood pressure in male patients with essential hypertension. Hypertension. 2004 Feb;43(2):192-7. doi: 10.1161/01.HYP.0000113293.15186.3b. Epub 2004 Jan 19. PMID 14732734
- [Background] Cagnacci A, Cannoletta M, Renzi A, Baldassari F, Arangino S, Volpe A. Prolonged melatonin administration decreases nocturnal blood pressure in women. Am J Hypertens. 2005 Dec;18(12 Pt 1):1614-8. doi: 10.1016/j.amjhyper.2005.05.008. PMID 16364834
- [Background] Grossman E, Laudon M, Yalcin R, Zengil H, Peleg E, Sharabi Y, Kamari Y, Shen-Orr Z, Zisapel N. Melatonin reduces night blood pressure in patients with nocturnal hypertension. Am J Med. 2006 Oct;119(10):898-902. doi: 10.1016/j.amjmed.2006.02.002. PMID 17000226
- [Background] Gubin DG, Gubin GD, Gapon LI, Weinert D. Daily Melatonin Administration Attenuates Age-Dependent Disturbances of Cardiovascular Rhythms. Curr Aging Sci. 2016;9(1):5-13. doi: 10.2174/1874609809666151130220011. PMID 26632428
- [Background] Mesri Alamdari N, Mahdavi R, Roshanravan N, Lotfi Yaghin N, Ostadrahimi AR, Faramarzi E. A double-blind, placebo-controlled trial related to the effects of melatonin on oxidative stress and inflammatory parameters of obese women. Horm Metab Res. 2015 Jun;47(7):504-8. doi: 10.1055/s-0034-1384587. Epub 2014 Aug 15. PMID 25126957
- [Background] Kozirog M, Poliwczak AR, Duchnowicz P, Koter-Michalak M, Sikora J, Broncel M. Melatonin treatment improves blood pressure, lipid profile, and parameters of oxidative stress in patients with metabolic syndrome. J Pineal Res. 2011 Apr;50(3):261-6. doi: 10.1111/j.1600-079X.2010.00835.x. Epub 2010 Dec 8. PMID 21138476
- [Background] Galley HF, Lowes DA, Allen L, Cameron G, Aucott LS, Webster NR. Melatonin as a potential therapy for sepsis: a phase I dose escalation study and an ex vivo whole blood model under conditions of sepsis. J Pineal Res. 2014 May;56(4):427-38. doi: 10.1111/jpi.12134. Epub 2014 Apr 5. PMID 24650045
- [Background] Lusardi P, Piazza E, Fogari R. Cardiovascular effects of melatonin in hypertensive patients well controlled by nifedipine: a 24-hour study. Br J Clin Pharmacol. 2000 May;49(5):423-7. doi: 10.1046/j.1365-2125.2000.00195.x. PMID 10792199
- [Background] Rechcinski T, Trzos E, Wierzbowska-Drabik K, Krzeminska-Pakula M, Kurpesa M. Melatonin for nondippers with coronary artery disease: assessment of blood pressure profile and heart rate variability. Hypertens Res. 2010 Jan;33(1):56-61. doi: 10.1038/hr.2009.174. Epub 2009 Oct 30. PMID 19876062
- [Background] Pickering TG, Hall JE, Appel LJ, Falkner BE, Graves JW, Hill MN, Jones DH, Kurtz T, Sheps SG, Roccella EJ; Council on High Blood Pressure Research Professional and Public Education Subcommittee, American Heart Association. Recommendations for blood pressure measurement in humans: an AHA scientific statement from the Council on High Blood Pressure Research Professional and Public Education Subcommittee. J Clin Hypertens (Greenwich). 2005 Feb;7(2):102-9. doi: 10.1111/j.1524-6175.2005.04377.x. No abstract available. PMID 15722655
- [Background] Fuchs SC, Poli-de-Figueiredo CE, Figueiredo Neto JA, Scala LC, Whelton PK, Mosele F, de Mello RB, Vilela-Martin JF, Moreira LB, Chaves H, Mota Gomes M, de Sousa MR, Silva RP, Castro I, Cesarino EJ, Jardim PC, Alves JG, Steffens AA, Brandao AA, Consolim-Colombo FM, de Alencastro PR, Neto AA, Nobrega AC, Franco RS, Sobral Filho DC, Bordignon A, Nobre F, Schlatter R, Gus M, Fuchs FC, Berwanger O, Fuchs FD. Effectiveness of Chlorthalidone Plus Amiloride for the Prevention of Hypertension: The PREVER-Prevention Randomized Clinical Trial. J Am Heart Assoc. 2016 Dec 13;5(12):e004248. doi: 10.1161/JAHA.116.004248. PMID 27965209
- [Background] Collier SR, Landram MJ. Treatment of prehypertension: lifestyle and/or medication. Vasc Health Risk Manag. 2012;8:613-9. doi: 10.2147/VHRM.S29138. Epub 2012 Nov 15. PMID 23172989
- [Result] Pandi-Perumal SR, BaHammam AS, Ojike NI, Akinseye OA, Kendzerska T, Buttoo K, Dhandapany PS, Brown GM, Cardinali DP. Melatonin and Human Cardiovascular Disease. J Cardiovasc Pharmacol Ther. 2017 Mar;22(2):122-132. doi: 10.1177/1074248416660622. Epub 2016 Jul 27. PMID 27450357
- [Result] Dominguez-Rodriguez A, Abreu-Gonzalez P, Reiter RJ. Melatonin and cardiovascular disease: myth or reality? Rev Esp Cardiol (Engl Ed). 2012 Mar;65(3):215-8. doi: 10.1016/j.recesp.2011.10.009. Epub 2012 Jan 13. No abstract available. English, Spanish. PMID 22245066

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/20/NCT03764020/Prot_SAP_000.pdf